CLINICAL TRIAL: NCT04841291
Title: Feasibility of Virtual Simulation-Based Diabetes Foot Care Education in Patients With Diabetes in Ethiopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fisseha Z Amdie (Other)
Responsible Party: Sponsor-Investigator, Fisseha Z Amdie, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 6032644
Record Dates: First submitted 2021-04-03; First posted 2021-04-12 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Foot Care
Keywords: Diabetes; Feasibility; Acceptability; Practicability; Foot-Care
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Access to virtual simulation-based diabetes foot care education for once for 30 minutes.
Who Masked: Outcomes Assessor
Masking Description: Data collectors will not be informed about participants' group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Simulation-Based Arm (Experimental): Access virtual simulation-based diabetes foot care education once for 30 minutes plus the standard care.
  Interventions: Behavioral: Diabetes Foot Care Education (DFCE)
- Standard Care Arm (No Intervention): Participants will continue utilizing the usual follow-up diabetes care which occurs every month.

INTERVENTIONS:
Behavioral: Diabetes Foot Care Education (DFCE) — Virtual simulation-based DFCE sessions on seven topics (the reasons for inspecting one's feet, risk factors and prevention strategies of diabetic foot ulcer, how to wash and moisturize feet, comfortable sock and shoe choices, what to look for, and what to do during feet inspection, how to trim fingernails, and how to maintain foot health) at University of Gondar computer lab for 30 minutes.
  Arms: Virtual Simulation-Based Arm

SUMMARY:
The primary aim of this study is to evaluate the feasibility of virtual simulation-based diabetes foot care education on foot care knowledge and practice/behaviour.

Research Questions

The primary question for this study is:

• Is virtual simulation-based diabetes foot care education a practical and acceptable intervention among patients with diabetes in Ethiopia?

The secondary questions are:

* What is the impact of virtual simulation-based diabetes foot care education on diabetes foot self-care knowledge among patients with diabetes mellitus?
* What is the impact of virtual simulation-based diabetes foot care education on diabetes foot self-care behaviour among patients with diabetes mellitus?
* What is the impact of virtual simulation-based diabetes foot care education on diabetes foot self-care efficacy among patients with diabetes mellitus?
* What is the impact of virtual simulation-based diabetes foot care education on diabetes foot health-belief among patients with diabetes mellitus?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years of age or older).
* Type II diabetes mellitus patients who are on diabetes follow-up at University of Gondar tertiary referral hospital

Exclusion Criteria:

* Patients with type 1 diabetes or gestational diabetes
* Patients who previously attended any form of formal Diabetes Self Management Education (DSME) program /documented/ in the past three months.
* Individuals with documented severe cognitive impairment
* Individuals with documented visual impairment that diminished their ability to navigate the game
* Terminally ill individuals
* Individuals without the ability to read or understand the Amharic consent documentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
The number of participants who accepted the virtual simulation-based foot care education. | One week after the commencement of intervention.
  Number of participants who scored 70 and above for the virtual simulation-based foot care education acceptance questionnaire.
The number of participants who believed in the practicality of the virtual simulation-based foot care education. | One week after the commencement of intervention.
  Number of participants who scored 70 and above for the virtual simulation-based foot care education practicality questionnaire.

SECONDARY OUTCOMES:
The participants' level of foot self-care knowledge. | Baseline and week one.
  Mean change from the baseline in foot self-care knowledge of participants one week after the commencement of the intervention. Diabetes foot self-care knowledge will be assessed with the Foot Care Knowledge (FCK) questionnaire. The Foot Care Knowledge questions evaluate the respondent's foot care knowledge. The maximum possible knowledge score will be 11 and can range from 1 to 11. A higher score means a better foot self-care knowledge.
The participants' level of foot self-care behavior. | Baseline and week one.
  Mean change from the baseline in foot self-care behavior of participants one week after the commencement of the intervention. Diabetes Foot Care Behavior will be assessed with the 15-item Foot Self-Care Behavior Scale (FSCBS). The Foot Self-Care Behavior Scale is a brief self-report questionnaire that measures foot care behavior. Patients will be asked to choose the most suitable response; never (1), rarely (2), sometimes (3), often (4), and always (5) to each question. The score ranged from 15-75 and a higher score indicates a better foot self-care behavior.
The participants' level of foot self-care efficacy to perform recommended diabetic foot self-care activities. | Baseline and week one.
  Mean change from the baseline in foot self-care efficacy of participants one week after the commencement of the intervention. This will be measured with Foot Care Confidence Scale (FCCS). The tool consists of 12 items on a 5-point Likert scale strongly not confident (1), not confident (2), moderately confident (3), confident (4), and strongly confident (5). The score ranged from 12 - 60; a higher score indicates a higher level of diabetes foot self-care efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Fisseha Zewdu Amdie, Msc., Principal Investigator — School of Nursing, Queen's University; Kevin Woo, Ph.D., Study Director — School of Nursing, Queen's University; Marian Luctkar-Flude, Ph.D., Study Director — School of Nursing, Queen's University; Erna Snelgrove-Clarke, Ph.D., Study Director — School of Nursing, Queen's University; Mona Sawhney, Ph.D., Study Director — School of Nursing, Queen's University
Locations (1):
- University of Gondar Referral Hospital, Gonder, Amhara, Ethiopia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abate TW, Enyew A, Gebrie F, Bayuh H. Nurses' knowledge and attitude towards diabetes foot care in Bahir Dar, North West Ethiopia. Heliyon. 2020 Nov 23;6(11):e05552. doi: 10.1016/j.heliyon.2020.e05552. eCollection 2020 Nov. PMID 33294694
- [Background] Aklilu T, Hiko D, Mohammed MA, Dekema NH. Diabetic Patients' Knowledge of Their Disease, Therapeutic Goals, and Self-management: Association With Goal Attainment at Dessie Referral Hospital, Ethiopia. Ther Innov Regul Sci. 2014 Sep;48(5):583-591. doi: 10.1177/2168479014524960. PMID 30231456
- [Background] Worku D, Hamza L, Woldemichael K. Patterns of diabetic complications at jimma university specialized hospital, southwest ethiopia. Ethiop J Health Sci. 2010 Mar;20(1):33-9. doi: 10.4314/ejhs.v20i1.69424. PMID 22434958
- [Background] Angamo MT, Melese BH, Ayen WY. Determinants of glycemic control among insulin treated diabetic patients in Southwest Ethiopia: hospital based cross sectional study. PLoS One. 2013 Apr 19;8(4):e61759. doi: 10.1371/journal.pone.0061759. Print 2013. PMID 23620789
- [Background] Aschalew AY, Yitayal M, Minyihun A, Bisetegn TA. Self-care practice and associated factors among patients with diabetes mellitus on follow up at University of Gondar Referral Hospital, Gondar, Northwest Ethiopia. BMC Res Notes. 2019 Sep 18;12(1):591. doi: 10.1186/s13104-019-4630-4. PMID 31533833
- [Background] Beran D, Yudkin JS. Diabetes care in sub-Saharan Africa. Lancet. 2006 Nov 11;368(9548):1689-95. doi: 10.1016/S0140-6736(06)69704-3. PMID 17098088
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Boren SA, Gunlock TL, Peeples MM, Krishna S. Computerized learning technologies for diabetes: a systematic review. J Diabetes Sci Technol. 2008 Jan;2(1):139-46. doi: 10.1177/193229680800200121. PMID 19885190
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Chali SW, Salih MH, Abate AT. Self-care practice and associated factors among Diabetes Mellitus patients on follow up in Benishangul Gumuz Regional State Public Hospitals, Western Ethiopia: a cross-sectional study. BMC Res Notes. 2018 Nov 26;11(1):833. doi: 10.1186/s13104-018-3939-8. PMID 30477553
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Dettori J. The random allocation process: two things you need to know. Evid Based Spine Care J. 2010 Dec;1(3):7-9. doi: 10.1055/s-0030-1267062. No abstract available. PMID 22956922
- [Background] Dube L, Van den Broucke S, Dhoore W, Kalweit K, Housiaux M. An Audit of Diabetes Self-Management Education Programs in South Africa. J Public Health Res. 2015 Nov 17;4(3):581. doi: 10.4081/jphr.2015.581. eCollection 2015 Nov 17. PMID 26753160
- [Background] Edelman SV. Taking Control Of Your Diabetes: An Innovative Approach to Improving Diabetes Care Through Educating, Motivating, and Making the Connection Between Patients and Health Care Providers. Clin Diabetes. 2017 Dec;35(5):333-339. doi: 10.2337/cd17-0090. No abstract available. PMID 29263578
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Embil JM, Albalawi Z, Bowering K, Trepman E. Foot Care. Can J Diabetes. 2018 Apr;42 Suppl 1:S222-S227. doi: 10.1016/j.jcjd.2017.10.020. No abstract available. PMID 29650101
- [Background] Foronda CL, Fernandez-Burgos M, Nadeau C, Kelley CN, Henry MN. Virtual Simulation in Nursing Education: A Systematic Review Spanning 1996 to 2018. Simul Healthc. 2020 Feb;15(1):46-54. doi: 10.1097/SIH.0000000000000411. PMID 32028447
- [Background] Gudina EK, Amade ST, Tesfamichael FA, Ram R. Assessment of quality of care given to diabetic patients at Jimma University Specialized Hospital diabetes follow-up clinic, Jimma, Ethiopia. BMC Endocr Disord. 2011 Dec 20;11:19. doi: 10.1186/1472-6823-11-19. PMID 22185229
- [Background] Indrayana S, Guo SE, Lin CL, Fang SY. Illness Perception as a Predictor of Foot Care Behavior Among People With Type 2 Diabetes Mellitus in Indonesia. J Transcult Nurs. 2019 Jan;30(1):17-25. doi: 10.1177/1043659618772347. Epub 2018 Apr 26. PMID 29699462
- [Background] Johnson C, Feenan K, Setliff G, Pereira K, Hassell N, Beresford HF, Epps S, Nicollerat J, Tatum W, Feinglos M, Vorderstrasse A. Building a Virtual Environment for Diabetes Self-Management Education and Support. Int J Virtual Communities Soc Netw. 2013;5(3):111359. doi: 10.4018/ijvcsn.2013070105. PMID 25699133
- [Background] Kasiya MM, Mang'anda GD, Heyes S, Kachapila R, Kaduya L, Chilamba J, Goodson P, Chalulu K, Allain TJ. The challenge of diabetic foot care: Review of the literature and experience at Queen Elizabeth Central Hospital in Blantyre, Malawi. Malawi Med J. 2017 Jun;29(2):218-223. doi: 10.4314/mmj.v29i2.26. No abstract available. PMID 28955436
- [Background] Lateef F. Simulation-based learning: Just like the real thing. J Emerg Trauma Shock. 2010 Oct;3(4):348-52. doi: 10.4103/0974-2700.70743. PMID 21063557
- [Background] Luctkar-Flude M, Tyerman J, Ziegler E, Carroll B, Shortall C, Chumbley L, Tregunno D. Developing a Sexual Orientation and Gender Identity Nursing Education Toolkit. J Contin Educ Nurs. 2020 Sep 1;51(9):412-419. doi: 10.3928/00220124-20200812-06. PMID 32833031
- [Background] McInnes A, Jeffcoate W, Vileikyte L, Game F, Lucas K, Higson N, Stuart L, Church A, Scanlan J, Anders J. Foot care education in patients with diabetes at low risk of complications: a consensus statement. Diabet Med. 2011 Feb;28(2):162-7. doi: 10.1111/j.1464-5491.2010.03206.x. PMID 21219423
- [Background] Petit dit Dariel OJ, Raby T, Ravaut F, Rothan-Tondeur M. Developing the Serious Games potential in nursing education. Nurse Educ Today. 2013 Dec;33(12):1569-75. doi: 10.1016/j.nedt.2012.12.014. Epub 2013 Jan 16. PMID 23332500
- [Background] Sari Y, Upoyo AS, Isworo A, Taufik A, Sumeru A, Anandari D, Sutrisna E. Foot self-care behavior and its predictors in diabetic patients in Indonesia. BMC Res Notes. 2020 Feb 1;13(1):38. doi: 10.1186/s13104-020-4903-y. PMID 32005281
- [Background] Torgerson DJ, Roberts C. Understanding controlled trials. Randomisation methods: concealment. BMJ. 1999 Aug 7;319(7206):375-6. doi: 10.1136/bmj.319.7206.375. No abstract available. PMID 10435967
- [Background] Verkuyl M, Hughes M, Tsui J, Betts L, St-Amant O, Lapum JL. Virtual Gaming Simulation in Nursing Education: A Focus Group Study. J Nurs Educ. 2017 May 1;56(5):274-280. doi: 10.3928/01484834-20170421-04. PMID 28467555
- [Background] Zhang Y, Liu C, Luo S, Xie Y, Liu F, Li X, Zhou Z. Factors Influencing Patients' Intentions to Use Diabetes Management Apps Based on an Extended Unified Theory of Acceptance and Use of Technology Model: Web-Based Survey. J Med Internet Res. 2019 Aug 13;21(8):e15023. doi: 10.2196/15023. PMID 31411146
- [Derived] Amdie FZ, Luctkar-Flude M, Snelgrove-Clarke E, Sawhney M, Alemu S, Woo K. Feasibility of Virtual Simulation-Based Diabetes Foot Care Education in Patients with Diabetes in Ethiopia: Protocol for a Randomized Controlled Trial. Diabetes Metab Syndr Obes. 2022 Mar 31;15:995-1009. doi: 10.2147/DMSO.S345722. eCollection 2022. PMID 35386589